CLINICAL TRIAL: NCT03141775
Title: Incidence and Economic Burden of Community and Hospital- Acquired Clostridium Difficile Infections (CDI) in the German Health Care System (IBIS)
Brief Title: Incidence and Economic Burden of Clostridium Difficile Infections (CDI) in the German Health Care System (IBIS)
Acronym: IBIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Maria J.G.T. Vehreschild, PD MD, University of Cologne
Other Study IDs: IBIS
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Clostridium Difficile Infection; Clostridium Difficile Diarrhea
Keywords: Clostridium difficile associated diarrhea (CDAD)
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment of CDI: Treatment of CDI for hospitalized patients with Clostridium difficile associated diarrhea
  Interventions: Other: Treatment of CDI

INTERVENTIONS:
Other: Treatment of CDI — Treatment (e.g. antibiotics, fecal microbiota transfer (FMT), probiotics) for patients with Clostridium difficile associated diarrhea

SUMMARY:
IBIS is a prospective, observational study, which aims to assess the cost of CDI per day, hospitalization and year including description of incremental costs in hospitalized patients, and recurrent episodes, in German hospitals. Exposure to CDI drugs will not be influenced and remains at the discretion of the treating physician.

In addition to treatment, Health-related quality of life (HRQL) will be analyzed using standardized questionnaires.

DETAILED DESCRIPTION:
Documentation of patient is performed by using the web-based survey platform www.ClinicalSurveys.net which was set up by researchers of the University Hospital of Cologne. This survey platform enables an optimal performance in epidemiological, observational, and interventional trials and is characterized by layered access security and frequent data backup. It has been used for numerous registry and cohort studies with approval of competent authorities and ethics boards.

The following two differences of data documentation are observed:

1. Retrospective data documentation:

   Data of patients that are too sick to provide informed consent, (up to 30% of all patients enrolled) will be obtained retrospectively, at least 90 days after diagnosis and will be documented in an anonymized fashion. For these patients, documentation of HRQL will not be feasible.
2. Prospective data documentation:

Data of patients with an informed consent.

The following data items are retrospectively or prospectively documented into our database, depending on if a informed consent exists or not:

* Demography: age (yrs), gender (m/f), comorbidities (as categories)
* Charlson Comorbidity Index (CCI)
* Karnofsky Score (0-100%)
* APACHE Score for patients in ICU
* Number of hospitalizations in the past 12 months prior to the CDI index episode
* Type and duration of antibiotic treatment during the last 3 months
* Diagnostic measures (microbiological tests, imaging, endoscopy) leading to diagnosis of CDI
* Severe and/or complicated CDI (Severe: white blood cell count ≥15 × 10³/μL and/or an increase in creatinine ≥1.5 times the baseline level; complicated: at least 1 of the following: hypotension requiring vasopressors, ICU admission for a complication of CDI, ileus leading to installation of a nasogastric tube, toxic megacolon, colonic perforation, or colectomy)
* Bowel movements: frequency and consistence according to Bristol stool scale (see appendix 1)
* Treatment for CDI: substance, dosage, frequency, duration
* Other antibiotic treatment: substance, dosage, frequency, duration
* Diagnosis of CDI recurrence: time point, diagnostic measures
* Treatment of CDI recurrence: substance, dosage, frequency, duration
* Duration of hospitalization: overall, types (general, intermediate care, intensive care, bone marrow transplantation)
* Mechanical ventilation (y/n)
* Days with contact isolation
* Days in single room
* Adverse drug reactions
* Health-related quality of life (HRQL) as determined by Garey et al. J Clin Gastroenterol 2016 (for prospective analysis only)

ELIGIBILITY:
Inclusion Criteria:

* Index episode of CDI based on

  * the presence of diarrhea (defined as ≥3 unformed bowel movements/24h) plus
  * an enzyme immunoassay (EIA) detecting Glutamate dehydrogenase (GDH) or polymerase chain reaction (PCR) for toxin B test plus
  * a positive EIA for toxin A and B
* Ongoing or new hospitalization at inclusion into the study.
* Written informed consent (IC) has been obtained from the study subject or a legal representative.

Exclusion Criteria:

* Patient with any social or logistical condition which in the opinion of the investigator may interfere with the conduct of the study, such as incapacity to well understand, not willing to collaborate, or cannot easily be contacted after discharge.
* CDI episode within the previous 84 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with a CDI episode in German hospitals
Sampling Method: Non-Probability Sample
Enrollment: 541 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of the cost of CDI index and recurrent episodes in German hospitals | 90 days
  Analyse direct and indirect costs associated with CDI per day, hospitalization and year including description of incremental costs in hospitalized patients.

SECONDARY OUTCOMES:
Assessment of health-related quality of life (HRQL) | 90 days
  Assessment of quality of life of patients with an CDI episode using a QoL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vehreschild, MD, Principal Investigator — University Hospital of Cologne, Department of Internal Medicine / Infectious Diseases, Cologne, Germany
Locations (6):
- Germany (6):
  - Städtisches Klinikum München, Munich, Bavaria
  - University Hospital Magdeburg, Magdeburg, Saxony-Anhalt
  - University Hospital Jena, Jena, Thuringia
  - University Hospital of Cologne, Cologne
  - Hospital Porz am Rhein, Cologne
  - University Clinical Center Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vehreschild MJ, Weitershagen D, Biehl LM, Tacke D, Waldschmidt D, Tox U, Wisplinghoff H, Von Bergwelt-Baildon M, Cornely OA, Vehreschild JJ. Clostridium difficile infection in patients with acute myelogenous leukemia and in patients undergoing allogeneic stem cell transplantation: epidemiology and risk factor analysis. Biol Blood Marrow Transplant. 2014 Jun;20(6):823-8. doi: 10.1016/j.bbmt.2014.02.022. Epub 2014 Mar 6. PMID 24607558
- [Background] Bauer MP, Notermans DW, van Benthem BH, Brazier JS, Wilcox MH, Rupnik M, Monnet DL, van Dissel JT, Kuijper EJ; ECDIS Study Group. Clostridium difficile infection in Europe: a hospital-based survey. Lancet. 2011 Jan 1;377(9759):63-73. doi: 10.1016/S0140-6736(10)61266-4. PMID 21084111
- [Background] Hensgens MP, Goorhuis A, Dekkers OM, van Benthem BH, Kuijper EJ. All-cause and disease-specific mortality in hospitalized patients with Clostridium difficile infection: a multicenter cohort study. Clin Infect Dis. 2013 Apr;56(8):1108-16. doi: 10.1093/cid/cis1209. Epub 2013 Jan 8. PMID 23300235